CLINICAL TRIAL: NCT02541708
Title: Intravenous Ferric Carboxymaltose Compared With Oral Iron in the Treatment of Iron Deficiency Anemia at Delivery in Tanzania
Brief Title: IV Ferric Carboxymaltose Compared With Oral Iron in the Treatment of Iron Deficiency Anemia at Delivery in Tanzania
Acronym: Ferinject
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ifakara Health Institute (Other)
Collaborators: Swiss Tropical & Public Health Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IFCIDA 001-2015
Record Dates: First submitted 2015-08-12; First posted 2015-09-04 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Iron-Deficiency Anemia
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — ferric carboxymaltose; ferrous sulfate; Folic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IV ferric carboxymaltose (Experimental): IV Ferric carboxymaltose is given at a dose calculated according to the severity of anemia and patients weight. The maximal weekly dose is 1000mg. If total dose exceeds 1000mg the dose is split in 1-3 infusions with one infusion per week.
  Interventions: Drug: Ferric carboxymaltose
- Ferrous sulphate 60mg+Folic acid 0.25mg (Active Comparator): Three dried ferrous sulphate and folic acid tablets every morning 30 mins before the meal. If side effects occur the drug may be taken with the meal or in 2 separate doses per day. The treatment will be pursued for 3 months after correction of anemia.
  Interventions: Drug: Ferrous sulfate + folic acid

INTERVENTIONS:
Drug: Ferric carboxymaltose — Intravenous Ferric carboxymaltose given at a calculated dose of 20mg/kg body weight in 1-3 infusions according to severity of anemia
  Other Names: Ferinject
  Arms: IV ferric carboxymaltose
Drug: Ferrous sulfate + folic acid — Three dried ferrous sulfate and folic acid tablets every morning 30 mins before the meal. If side effects occur the drug may be taken with the meal or in 2 separate doses per day. The treatment will be pursued for 3 months after correction of anemia
  Other Names: Fefo
  Arms: Ferrous sulphate 60mg+Folic acid 0.25mg

SUMMARY:
Intravenous iron preparations have been shown to be superior to oral iron and have largely replaced the treatment of anaemia in Northern countries. However, the socio-economic and medical conditions in low resource countries greatly differ from those in northern countries. Patients' different access to medication supply, perception of medication need and compliance as well as the burden of concomitant disease like malaria, soil-transmitted helminths, schistosomiasis, HIV and red blood cells (RBC) genetic disorders may influence effectiveness and safety of iron substitution modality. The aim of the present study is to compare iv iron substitution by ferric carboxymaltose (Ferinject®) to per oral iron substitution in a low resource country

DETAILED DESCRIPTION:
The objectives of the study are as follows:

Primary objective:

To assess the superiority in terms of effectiveness of iv iron substitution with ferric carboxymaltose versus per oral iron substitution in women with iron deficient anemia at delivery in Tanzania.

Secondary objectives

* To evaluate safety and feasibility of intravenous ferric carboxymaltose substitution compared to per oral iron substitution in a resource limited country
* To evaluate acceptance of intravenous ferric carboxymaltose substitution compared to per oral iron substitution in a resource limited country
* To evaluate wellbeing of women receiving intravenous ferric carboxymaltose compared to women receiving per oral iron substitution
* To evaluate the sensitivity of diagnosis of iron deficiency by measuring hemoglobin, mean corpuscular volume (MCV) and mean corpuscular hemoglobin concentration (MCHC) only, compared to the diagnosis by measuring iron metabolism parameters in a resource limited country

ELIGIBILITY:
Inclusion Criteria:

* Women close to delivery
* Screening will be performed using the HemoCue System. In case of anemia, defined by Hg <110 g/l, a venous puncture will be performed and the blood analyzed on a 5 population analyzer with erythrocyte indices and Reticulocyte indices and ferritin determined. Then If the anemia defined as Hg <110 g/l is confirmed and the if ferritin is below 50 ng/ml, the patient will be included in the present study
* Patient compliance and geographic proximity allow proper staging and follow-up
* Patient must give written informed consent before registration

Exclusion Criteria:

* Active malaria; patients will be tested for malaria by Rapid Diagnostic Test and microscopy and if positive treated. Patient with treated malaria can be included
* Helminthic infection; patients will be tested for helminthic infections by a stool ova and parasite exam and if positive treated by single oral dose of 400 mg albendazole. Treated patients can be included.
* HIV positivity. Patients will be tested and if positive they will be referred to the Care and Treatment Clinic at Bagamoyo District Hospital and excluded from the study.
* Known hemoglobinopathy
* C-Reactive protein (CRP) >20
* Patients with chronic fever
* Psychiatric disorder precluding understanding of information on trial related topics or giving informed consent
* Concurrent treatment with other experimental drugs or treatment in another clinical trial within 30 days prior to trial entry
* Any serious underlying medical condition (at the judgment of the investigator) which could impair the ability of the patient to participate in the trial
* Known allergy or hypersensitivity to study drug.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 230 (Actual)
Dates: Start 2015-09; Primary Completion 2018-04 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Percentage of women with correction of hemoglobin to normal values (Hb> 11.5g/dl) at 6 weeks by treatment arm | 6 weeks
  The proportion of women in each trial arm who have attained the corrected hemoglobin to normal values after starting trial treatment.

SECONDARY OUTCOMES:
Best response (Hemoglobin) in grams per decilitre (g/dl) | up to 1 year
  Is the highest hemoglobin value or maximal hemoglobin increase after start of study medication
Percentage of women with corrected iron deficiency (Ferritin>50ng/ml) in each arm | 6 weeks
  The proportion of women in each trial arm who have attained the corrected serum ferritin levels to normal values after starting trial treatment in nanograms per milliltre(ng/mL)
Best response (Ferritin) in nanograms per milliltre (ng/mL) | up to 1 year
  Is the highest ferritin value or maximal ferritin increase after start of study medication.
  The proportion of women in each trial arm who have attained the corrected serum ferritin levels to normal values after starting trial treatment
Time to response (Hemoglobin) in weeks | up to 1 year
  Is the time interval between the date of start of study medication until the date of reaching maximal hemoglobin value
Time to response (Ferritin) in weeks | up to 1 year
  Is the time interval between the date of start of study medication until the date of reaching maximal ferritin value
Response duration (Hemoglobin) in weeks | up to 1 year
  Is the time from the date when the highest hemoglobin value is reached until the date of decrease to Hb<11.5 g/dl or a decrease of more than 1 g/dl
Response duration (Ferritin) in weeks | up to 1 year
  Is the time from the date when the highest ferritin value is reached until the date of decrease to ferritin<50 ng/ml
Frequency and severity of solicited and non-solicited adverse events after IV ferric carboxymaltose substitution and oral iron substitution | up to 1 year
  Number of participants with adverse events either clinical events or abnormal laboratory values with grading of severity reported according to the Common Terminology Criteria of Adverse Events (CTCAE) version 4
Compliance to study medication intake after intravenous ferric carboxymaltose substitution and oral iron substitution (Questionnaire and pill count) | up to 1 year
  The proportion of women in each trial arm who have completed the trial related treatment either the number of prescribed infusions of ferric carboxymaltose or oral tablets of ferrous sulphate and folic acid

OTHER OUTCOMES:
Sensitivity of erythrocyte indices for the diagnosis of iron deficiency anemia in Tanzania (parameters used are mean corpuscular volume(MCV) and mean corpuscular hemoglobin concentration(MCHC) | 1 year
  Is the probability that a test (erythrocyte indices) will indicate iron deficiency among participants with the disease as confirmed by iron metabolism parameters (Gold standard). It will be reported as percentage.
Specificity of erythrocyte indices for the diagnosis of iron deficiency anemia in Tanzania ((parameters used are mean corpuscular volume(MCV) and mean corpuscular hemoglobin concentration(MCHC) | 1 year
  Is the fraction of those without disease (iron deficiency) confirmed by iron metabolism parameters who will have a negative test (erythrocyte indices) results. It will be reported as percentage.
Positive predictive value of erythrocyte indices for the diagnosis of iron deficiency anemia in Tanzania (parameters used are mean corpuscular volume(MCV) and mean corpuscular hemoglobin concentration(MCHC) | 1 year
  Is the proportion of participants who truly have the disease(iron deficiency) as confirmed by iron metabolism parameters among the total number of participants with positive test results(erythrocyte indices). It will be reported as percentage.
Negative predictive value of erythrocyte indices for the diagnosis of iron deficiency anemia in Tanzania (parameters used are mean corpuscular volume(MCV) and mean corpuscular hemoglobin concentration(MCHC) | 1 year
  Is the proportion of participants who do not have the disease(iron deficiency) as confirmed by iron metabolism parameters among the total number of participants with negative test results(erythrocyte indices). It will be reported as percentage.

CONTACTS AND LOCATIONS:
Overall Officials: Sandrine Meyer-Monard, PD DrMed, Principal Investigator — Swiss Tropical & Public Health Institute; Salim Abdulla, MD,PhD, Study Chair — Ifakara Health Institute; Marcel Tanner, PhD, MPH, Study Chair — Swiss Tropical & Public Health Institute
Locations (1):
- Ifakara Health Institute, Bagamoyo, Tanzania

REFERENCES:
- [Background] van Hensbroek MB, Jonker F, Bates I. Severe acquired anaemia in Africa: new concepts. Br J Haematol. 2011 Sep;154(6):690-5. doi: 10.1111/j.1365-2141.2011.08761.x. Epub 2011 Jun 28. PMID 21707575
- [Background] Balarajan Y, Ramakrishnan U, Ozaltin E, Shankar AH, Subramanian SV. Anaemia in low-income and middle-income countries. Lancet. 2011 Dec 17;378(9809):2123-35. doi: 10.1016/S0140-6736(10)62304-5. Epub 2011 Aug 1. PMID 21813172
- [Background] Bodnar LM, Scanlon KS, Freedman DS, Siega-Riz AM, Cogswell ME. High prevalence of postpartum anemia among low-income women in the United States. Am J Obstet Gynecol. 2001 Aug;185(2):438-43. doi: 10.1067/mob.2001.115996. PMID 11518906
- [Background] Zimmermann MB, Chassard C, Rohner F, N'goran EK, Nindjin C, Dostal A, Utzinger J, Ghattas H, Lacroix C, Hurrell RF. The effects of iron fortification on the gut microbiota in African children: a randomized controlled trial in Cote d'Ivoire. Am J Clin Nutr. 2010 Dec;92(6):1406-15. doi: 10.3945/ajcn.110.004564. Epub 2010 Oct 20. PMID 20962160
- [Background] Lynch SR. Why nutritional iron deficiency persists as a worldwide problem. J Nutr. 2011 Apr 1;141(4):763S-768S. doi: 10.3945/jn.110.130609. Epub 2011 Mar 2. PMID 21367937
- [Background] Van Wyck DB, Martens MG, Seid MH, Baker JB, Mangione A. Intravenous ferric carboxymaltose compared with oral iron in the treatment of postpartum anemia: a randomized controlled trial. Obstet Gynecol. 2007 Aug;110(2 Pt 1):267-78. doi: 10.1097/01.AOG.0000275286.03283.18. PMID 17666600
- [Background] Van Wyck DB, Mangione A, Morrison J, Hadley PE, Jehle JA, Goodnough LT. Large-dose intravenous ferric carboxymaltose injection for iron deficiency anemia in heavy uterine bleeding: a randomized, controlled trial. Transfusion. 2009 Dec;49(12):2719-28. doi: 10.1111/j.1537-2995.2009.02327.x. Epub 2009 Jul 22. PMID 19682342
- [Background] Moore RA, Gaskell H, Rose P, Allan J. Meta-analysis of efficacy and safety of intravenous ferric carboxymaltose (Ferinject) from clinical trial reports and published trial data. BMC Blood Disord. 2011 Sep 24;11:4. doi: 10.1186/1471-2326-11-4. PMID 21942989
- [Background] Rohner F, Zimmermann MB, Amon RJ, Vounatsou P, Tschannen AB, N'goran EK, Nindjin C, Cacou MC, Te-Bonle MD, Aka H, Sess DE, Utzinger J, Hurrell RF. In a randomized controlled trial of iron fortification, anthelmintic treatment, and intermittent preventive treatment of malaria for anemia control in Ivorian children, only anthelmintic treatment shows modest benefit. J Nutr. 2010 Mar;140(3):635-41. doi: 10.3945/jn.109.114256. Epub 2010 Jan 27. PMID 20107144
- [Background] Beard JL, Hendricks MK, Perez EM, Murray-Kolb LE, Berg A, Vernon-Feagans L, Irlam J, Isaacs W, Sive A, Tomlinson M. Maternal iron deficiency anemia affects postpartum emotions and cognition. J Nutr. 2005 Feb;135(2):267-72. doi: 10.1093/jn/135.2.267. PMID 15671224
- [Derived] Vanobberghen F, Lweno O, Kuemmerle A, Mwebi KD, Asilia P, Issa A, Simon B, Mswata S, Schmidlin S, Glass TR, Abdulla S, Daubenberger C, Tanner M, Meyer-Monard S. Efficacy and safety of intravenous ferric carboxymaltose compared with oral iron for the treatment of iron deficiency anaemia in women after childbirth in Tanzania: a parallel-group, open-label, randomised controlled phase 3 trial. Lancet Glob Health. 2021 Feb;9(2):e189-e198. doi: 10.1016/S2214-109X(20)30448-4. Epub 2020 Nov 24. PMID 33245866
- See also: Swiss Tropical and Public Health Institute — http://www.swisstph.ch
- See also: Ifakara Health Institute — http://www.ihi.or.tz
- See also: National Institute for Medical Research — http://www.nimr.or.tz